CLINICAL TRIAL: NCT07026383
Title: Physiological and Psychological Profiles of the Athletic Women and the Risk of Sport Injuries in Saudi Arabia
Brief Title: Physiological and Psychological Profiles
Status: Recruiting | Type: Observational
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, PNU, Princess Nourah Bint Abdulrahman University
Other Study IDs: PNU-4
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer; Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- athletic
  Interventions: Behavioral: performance test

INTERVENTIONS:
Behavioral: performance test — Injury risk was evaluated using the Lower Extremity Functional Test (LEFT), which involves eight agility drills performed consecutively on a diamond-shaped course without rest intervals. The test includes eight components-forward run, backward run, side shuffle, carioca, figure-eight run, 45-degree cuts, 90-degree cuts, and a counter vertical jump-along with the single-leg hop for distance, following a standardized testing protocol known to predict injury risk. Participants who took longer to complete the test were categorized into the high injury risk group, while those with shorter completion times were classified into the low injury risk group.

SUMMARY:
The participation of women in high-impact sports such as rugby and basketball has been steadily increasing in Saudi Arabia. These sports are known for their physical demands and competitive nature, which have heightened the incidence of sports-related injuries. Understanding the predictive factors for these injuries is critical for developing preventive strategies, reducing long-term health consequences, and reducing healthcare burdens. Therefore, this study aims to identify the predictive effect of physiological factors (e.g., muscle strength, anaerobic power, oxygen consumption) and psychological factors (e.g., self-efficacy, resilience) on sports injuries among female athletes in Saudi Arabia, particularly focusing on those involved in rugby and basketball.

A prospective cross-sectional design will be employed, involving a total of 30 female athletes aged 18-35 years actively participating in rugby and basketball. Data will be collected at the lifestyle research center through a series of physiological assessments, including maximal oxygen consumption, anaerobic power testing, isokinetic muscle strength testing, and psychological evaluations using validated questionnaires. The findings are expected to provide insights into the specific factors that increase injury risk among Saudi female athletes, offering targeted strategies for injury prevention. These strategies aim not only to minimize injuries but also to reduce associated healthcare costs, thereby supporting the sustainable growth of women's sports in Saudi Arabia. Ultimately, this study seeks to contribute to the broader objectives of Vision 2030 by promoting a vibrant sports culture and enhancing public health.

ELIGIBILITY:
Inclusion Criteria:

* Female athletes aged 18-35 years recruited from rugby and basketball teams in Saudi Arabia
* Actively involved in rugby and basketball
* Minimum of one year of experience in their respective sport
* Regular participation in training and competitive events

Exclusion Criteria:

* Recent injury within the last six months that limits athletic performance Pregnancy
* Presence of any chronic medical condition that could influence study outcomes
* Uncontrolled diabetes or hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study participants will be selected from female athletes aged 18 to 35 years who are actively participating in rugby and basketball teams in Saudi Arabia. These athletes are involved in regular training and competitive matches, have at least one year of experience in their respective sports, and represent the population of active female sports enthusiasts within this age group in the region.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption test: | baseline
  subjects will complete symptom limited treadmill exercise tests using a modification of Balkes protocol, which has been previously used among individuals with obesity. Participants will be connected to a gas analyzing metabolic cart (mouthpiece) for the determination of oxygen uptake, ventilated carbon dioxide, lung volumes, and heart rate through a gas analysis system using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) and HR monitor (Polar H7, Kempele, Finland).The tests will be performed on a computerized treadmill allowing programmed adjustment of both speed and inclination components of the work rate. The gas exchange system measured the oxygen consumption (VO2) and carbon dioxide production (VCO2) throughout the test.
Wingate test | baseline
  The Wingate test will be performed on a cycle ergometer (Ergomedic 828E, Monark, Sweden). Participants will perform a 30-second all-out sprint against a resistance equivalent to 7.5% of their body weight. The test measures the peak power (in watts), average power, and rate of fatigue. These metrics provide insights into the anaerobic performance capabilities of athletes.
Isokinetic muscle strength | baseline
  testing will be conducted using an isokinetic dynamometer (Humac Norm Isokinetic Software System-USA. The participants will perform knee flexion and extension at angular velocities of 60°/s and 180°/s. The peak torque (Nm) will be recorded for each movement, which indicates the maximum strength of the quadriceps and hamstrings. Bilateral comparisons will be performed to assess muscle imbalances, which are potential injury risk factors. Quadriceps and hamstring muscles of the dominant leg will be also examined. The dominant lower extremity was defined as the preferred leg for kicking the ball. The researcher will use a moderate pace and load (50-100 W), followed by 10 min of dynamic stretching concentrating on the lower limbs to prepare every participant for the assessment of leg torque.
The General Self-Efficacy Scale (GSES) | baseline
  The GSES is a self-report and unidimensional measure consisting of 10 items (e.g., "I can always manage to solve difficult problems if I try hard enough"). The total score ranges from 10 to 40, with higher scores indicating stronger belief that one's actions are responsible for successful outcomes.
Brief Resilience Scale (BRS) | baseline
  Brief Resilience Scale (BRS) is a self-rated assessment developed to quantify people's ability to bounce back and cope in accordance to health-related stressors.The overarch objective of this test was to provide the ability to thrive in the face of adversity. In other words, those who are more resilient are better able to cope with life challenges. The BRS was first developed by Smith et al.. and was used in this study. It comprises a six-item scale, with total possible points ranging from to 6-30. Each item has possible responses ranging from1= strongly disagree, 2= disagree, 3= neutral, 4= agree, and 5= Strongly Agree. The validity and reliability for this scale has been examined, giving excellent psychometric properties that allows for efficient measurement of resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- PNU, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided